CLINICAL TRIAL: NCT03727750
Title: A SINGLE ARM, OPEN-LABEL, PHASE 4 STUDY EVALUATING QT INTERVAL, PHARMACOKINETICS, AND SAFETY OF GEMTUZUMAB OZOGAMICIN (MYLOTARG (TRADEMARKER)) AS A SINGLE-AGENT REGIMEN IN PATIENTS WITH RELAPSED OR REFRACTORY CD33-POSITIVE ACUTE MYELOID LEUKEMIA
Brief Title: Evaluating QTc, PK, Safety of Gemtuzumab Ozogamicin (GO) in Patients With CD33+ R/R AML
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1761031; 2018-002619-89 (EudraCT Number)
Record Dates: First submitted 2018-09-28; First posted 2018-11-01 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-02

CONDITIONS: ECG; Pharmacokinetics; Safety
Keywords: gemtuzumab ozogamicin; Mylotarg; QT interval prolongation; Pharmacokinetics; Safety; Veno-occlusive disease; Anti-drug antibody
MeSH Terms: interventions — Gemtuzumab

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, interventional
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemtuzumab Ozogamicin (GO) (Experimental): Patients will receive three doses of Gemtuzumab Ozogamicin (GO) 3 mg/m2 (up to one vial) as a 2 hour intravenous infusion on Cycle 1 Days 1, 4, and 7. A second cycle of GO 3mg/m² (up to one vial) on Cycle 2 Days 1, 4, and 7 will be allowed at the investigator's discretion for patients who meet the criteria
  Interventions: Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Three doses of GO 3 mg/m2 (up to one vial) as a 2 hour intravenous infusion on Cycle 1 Days 1, 4, and 7. A second cycle of GO 3mg/m² (up to one vial) on Cycle 2 Days 1, 4, and 7 will be allowed at the investigator's discretion for patients who meet the criteria

SUMMARY:
This is a single-arm, open-label, Phase 4 study evaluating the effect of GO on the QTc, pharmacokinetics, safety, and immunogenicity of GO as a single-agent monotherapy in adult and pediatric patients with relapsed or refractory CD33-positive AML.

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase 4 study evaluating the effect of GO on the QTc, pharmacokinetics, safety, and immunogenicity of GO as a single-agent monotherapy in adult and pediatric patients with relapsed or refractory CD33-positive AML. Approximately 50 adult (age >=18 years) and 6 pediatric (12 years =< age =< 17 years) patients who satisfy the study eligibility criteria will be enrolled. Enrolled patients will receive GO 3 mg/m2 up to 2 cycles on Days 1, 4, and 7 at each cycle. The impact of GO on VOD/SOS in the context of previous and subsequent HSCT will also be assessed. Patients enrolled in the study will receive three doses of GO 3 mg/m2 (up to one vial) as a 2-hour intravenous infusion on Cycle 1 Days 1, 4, and 7. A second cycle of GO 3mg/m² (up to one vial) on Cycle 2 Days 1, 4, and 7 will be allowed at the investigator's discretion for patients who meet the following criteria after Cycle 1: Bone marrow with a decrease of blast percentage to at least 25% or a decrease of pretreatment blast percentage by at least 50%; and Blood count with neutrophils >=1,000/µL, and platelets >=50,000/µL, except in patients with the bone marrow blasts >=5%, the decrease in neutrophils and platelets thought to be due to the underlying leukemia. After GO treatment, subsequent anticancer therapy such as consolidation or conditioning regimen and/or HSCT could be considered at the investigator's discretion. A minimum interval of 2 months is recommended between the last dose of GO and HSCT.

ELIGIBILITY:
Inclusion Criteria

* Refractory or relapsed (ie, bone marrow blasts >5%) CD33-positive AML.
* Age >=12 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2.
* Initial peripheral white blood cells (WBC) counts >=30,000/mL; patients with a higher WBC count should undergo cytoreduction.
* Adequate renal/hepatic functions

Exclusion Criteria

* Patients with prior treatment with gemtuzumab ozogamicin (GO).
* Patients with prior history of VOD/SOS.
* Prior HSCT is not allowed, if it was conducted within 2 months prior to study enrollment.
* Patients with known active central nervous system (CNS) leukemia.
* Uncontrolled or active infectious status.
* Uncontrolled cardiac dysrhythmias of NCI CTCAE Grade 2, uncontrolled atrial fibrillation of any grade.
* Sero-positivity to human immunodeficieny virus (HIV).
* Active hepatitis B or hepatitis C infection
* Chemotherapy, radiotherapy, or other anti-cancer therapy (except hydroxyurea as cytoreduction) within 2 weeks prior to enrollment in the study.
* Major surgery within 4 weeks prior to enrollment.
* QTc interval >470 milliseconds (msec) using the Fridericia (QTcF), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
* The use of medications known to predispose to Torsades de Pointes within 2 weeks prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemtuzumab ozogamicin (GO).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (4):
  - Augusta University Medical Center Clinical Research Pharmacy, Augusta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - Research Transition Facility, Edmonton, Alberta
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Hamilton Health Sciences, Juravinski Hospital, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
- Hungary (4):
  - Semmelweis Egyetem I.sz Belgyogyaszati Klinika, Hematologiai Osztaly, Budapest
  - Debreceni Egyetem Klinikai Kozpont Belgyogyaszati Klinika, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, II. Belgyogyaszat - Hematologiai Osztaly, Győr
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
- Poland (4):
  - Klinika Hematologii i Transplantologii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku, Wroclaw
  - Pracownia Tomografii Komputerowej i Pracownia Rezonansu Magnetycznego, Wroclaw
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (3):
  - The Royal Bournemouth and Christchurch NHS Foundation Trust, Bournemouth, Dorset
  - Belfast Health and Social Care Trust, Belfast
  - Clatterbridge Cancer Center NHS Foundation Trust, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Montesinos P, Kota V, Brandwein J, Bousset P, Benner RJ, Vandendries E, Chen Y, McMullin MF. A phase IV study evaluating QT interval, pharmacokinetics, and safety following fractionated dosing of gemtuzumab ozogamicin in patients with relapsed/refractory CD33-positive acute myeloid leukemia. Cancer Chemother Pharmacol. 2023 May;91(5):441-446. doi: 10.1007/s00280-023-04516-9. Epub 2023 Mar 9. PMID 36892676
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1761031

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 66 participants signed the informed consent form and were screened. Out of 66 participants, 15 participants were screen failed and 51 participants were enrolled into the study
Groups:
- Gemtuzumab Ozogamicin (GO): Participants with confirmed diagnosis of refractory or relapsed cluster of differentiation (CD33)- positive Acute Myeloid Leukemia (AML) aged greater than or equal to (>=) 18 years received three doses of Gemtuzumab Ozogamicin, 3 milligram per meter square (mg/m^2) as intravenous (IV) infusion on Days 1, 4 and 7 of Cycle 1 and 2.
Period: Overall Study
Arm/Group | Gemtuzumab Ozogamicin (GO)
Started | 51
Safety Set | 50
Completed | 2
Not Completed | 49
Not completed — Death | 45
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all enrolled participants included in the study.
Groups:
- Gemtuzumab Ozogamicin (GO): Participants with confirmed diagnosis of refractory or relapsed CD33-positive Acute Myeloid Leukemia (AML) aged >= 18 years received three doses of Gemtuzumab Ozogamicin, 3 mg/m^2 as IV infusion on Days 1, 4 and 7 of Cycle 1 and 2.
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 39
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 1: 1 Hour
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. QT interval was the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle. QTcF was the QT interval corrected for heart rate using Fridericia's formula: QTcF = QT divided by cube root of 60/heart rate. Change from baseline in QT interval corrected for heart rate using Fridericia's formula was reported.
Time Frame: Baseline, Cycle 1 Day 1: 1 Hour
Population: QTc analysis set included all the participants in the safety analysis set who had a baseline ECG and at least 1 post-dose ECG. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 48
milliseconds | 4.90 [2.48 to 7.32]

2. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 1: 2 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 1 Day 1: 2 Hours
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 46
milliseconds | 4.25 [1.66 to 6.84]

3. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 1: 4 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 1 Day 1: 4 Hours
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 49
milliseconds | 5.10 [2.15 to 8.06]

4. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 4: 0 Hour
Description: as for outcome 1
Time Frame: Baseline, Cycle 1 Day 4: 0 Hour
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 47
milliseconds | -2.44 [-5.98 to 1.09]

5. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 4: 2 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 1 Day 4: 2 Hours
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 46
milliseconds | -0.45 [-3.98 to 3.07]

6. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 7: 0 Hour
Description: as for outcome 1
Time Frame: Baseline, Cycle 1 Day 7: 0 Hour
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 44
milliseconds | -1.00 [-4.59 to 2.58]

7. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 7: 2 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 1 Day 7: 2 Hours
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 45
milliseconds | 4.29 [0.88 to 7.70]

8. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 7: 4 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 1 Day 7: 4 Hours
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 44
milliseconds | 4.19 [0.45 to 7.93]

9. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 1 Day 7: 6 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 1 Day 7: 6 Hours
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 45
milliseconds | 1.03 [-2.88 to 4.93]

10. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 2 Day 1: 0 Hour
Description: as for outcome 1
Time Frame: Baseline, Cycle 2 Day 1: 0 Hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 9
milliseconds | 4.0 (11.32)

11. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 2 Day 1: 2 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 2 Day 1: 2 Hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 9
milliseconds | 7.3 (9.12)

12. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 2 Day 7: 0 Hour
Description: as for outcome 1
Time Frame: Baseline, Cycle 2 Day 7: 0 Hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 9
milliseconds | -5.4 (7.58)

13. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 2 Day 7: 2 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 2 Day 7: 2 Hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 9
milliseconds | -1.6 (10.69)

14. Primary Outcome: Change From Baseline in Corrected QT Interval for Heart Rate Using Fridericia's Formula (QTcF) at Cycle 2 Day 7: 6 Hours
Description: as for outcome 1
Time Frame: Baseline, Cycle 2 Day 7: 6 Hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 9
milliseconds | -8.8 (14.43)

15. Secondary Outcome: Clearance (CL) of Gemtuzumab Ozogamicin
Description: Clearance of a drug was measure of the rate at which the drug was metabolized or eliminated by normal biological processes.
Time Frame: Pre dose, 2, 4, 6, 72, 192 and 336 hours post dose on Cycle 1 Day 7
Population: Pharmacokinetic (PK) analysis set included all the participants who were treated with GO and contributed at least 1 PK sample. Here, 'Number Analyzed' = participants evaluable for this outcome measure for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
Liters/hour
  AC-CL-184538: number analyzed (Participants) | 47
  AC-CL-184538 | 15.02 (112)
  CL-184538: number analyzed (Participants) | 45
  CL-184538 | 4246 (177)
  Total HP67.6 Antibody: number analyzed (Participants) | 47
  Total HP67.6 Antibody | 0.3212 (153)

16. Secondary Outcome: Volume of Distribution of Gemtuzumab Ozogamicin
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: Pre dose, 2, 4, 6, 72, 192 and 336 hours post dose on Cycle 1 Day 7
Population: This outcome measure could not be estimated due to insufficient concentration-time data by non-compartmental analysis.
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 0

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): AC-CL-184538 and CL-184538
Description: Cmax was defined as the maximum observed plasma concentration of GO. Calicheamicin (conjugated calicheamicin ac-CL-184538 and unconjugated CL-184538) analyte were used to determined the Cmax in this outcome measure.
Time Frame: Pre dose, 1, 2, 4, 6, 24 and 72 hours post dose on Cycle 1 Day 1; and Pre dose, 2, 4, 6, 72, 192 and 336 hours post dose on Cycle 1 Day 7
Population: PK analysis set included all the participants who were treated with GO and contributed at least 1 PK sample. Here, 'Number Analyzed' = participants evaluable for this outcome measure for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/milliliter
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
picogram/milliliter
  Cycle 1 Day 1: AC-CL-184538 | 6457 (81)
  Cycle 1 Day 1: CL-184538 | 45.69 (51)
  Cycle 1 Day 7: AC-CL-184538: number analyzed (Participants) | 47
  Cycle 1 Day 7: AC-CL-184538 | 11740 (79)
  Cycle 1 Day 7: CL-184538: number analyzed (Participants) | 47
  Cycle 1 Day 7: CL-184538 | 58.76 (70)

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): Total HP67.6 Antibody
Description: Cmax was defined as the maximum observed plasma concentration of GO. Total HP67.6 antibodies analyte was used to determined the Cmax in this outcome measure.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
nanogram/milliliter
  Cycle 1 Day 1: Total HP67.6 Antibody | 282.1 (77)
  Cycle 1 Day 7: Total HP67.6 Antibody: number analyzed (Participants) | 47
  Cycle 1 Day 7: Total HP67.6 Antibody | 585.6 (105)

19. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax = time (hours) to maximum plasma concentration (Cmax).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
hours
  Cycle 1 Day 1: AC-CL-184538 | 2.080 [0.933 to 5.83]
  Cycle 1 Day 1: CL-184538: number analyzed (Participants) | 41
  Cycle 1 Day 1: CL-184538 | 2.170 [1.00 to 6.08]
  Cycle 1 Day 1: Total HP67.6 Antibody: number analyzed (Participants) | 49
  Cycle 1 Day 1: Total HP67.6 Antibody | 2.080 [0.933 to 4.25]
  Cycle 1 Day 7: AC-CL-184538: number analyzed (Participants) | 47
  Cycle 1 Day 7: AC-CL-184538 | 2.130 [0.000 to 6.25]
  Cycle 1 Day 7: CL-184538: number analyzed (Participants) | 45
  Cycle 1 Day 7: CL-184538 | 3.920 [1.85 to 6.10]
  Cycle 1 Day 7: Total HP67.6 Antibody: number analyzed (Participants) | 47
  Cycle 1 Day 7: Total HP67.6 Antibody | 2.170 [1.92 to 6.40]

20. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of Last Quantifiable Concentration (AUClast): AC-CL-184538 and CL-184538
Description: Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUClast). Calicheamicin (conjugated calicheamicin ac-CL-184538 and unconjugated CL-184538) analytes were used to determined the AUClast in this outcome measure.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/milliliter
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
picogram*hour/milliliter
  Cycle 1 Day 1: AC-CL-184538 | 93260 (83)
  Cycle 1 Day 1: CL-184538 | 99.83 (171)
  Cycle 1 Day 7: AC-CL-184538: number analyzed (Participants) | 47
  Cycle 1 Day 7: AC-CL-184538 | 453900 (120)
  Cycle 1 Day 7: CL-184538: number analyzed (Participants) | 47
  Cycle 1 Day 7: CL-184538 | 242.0 (283)

21. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of Last Quantifiable Concentration (AUClast): Total HP67.6 Antibody
Description: Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUClast). Total HP67.6 antibodies analyte was used to determined the AUClast in this outcome measure.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
nanogram*hour/milliliter
  Cycle 1 Day 1: Total HP67.6 Antibody | 2496 (210)
  Cycle 1 Day 7: Total HP67.6 Antibody: number analyzed (Participants) | 47
  Cycle 1 Day 7: Total HP67.6 Antibody | 14740 (388)

22. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time 72 Hours (AUC0-72): AC-CL-184538 and CL-184538
Description: Area under the plasma concentration-time curve from time zero to the time 72 hours (AUC0-72). Calicheamicin (conjugated calicheamicin ac-CL-184538 and unconjugated CL-184538) analytes were used to determined the AUC0-72 in this outcome measure.
Time Frame: Pre dose, 1, 2, 4, 6, 24 and 72 hours post dose on Cycle 1 Day 1
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/milliliter
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
picogram*hour/milliliter
  AC-CL-184538 | 93490 (82)
  CL-184538: number analyzed (Participants) | 36
  CL-184538 | 247.8 (176)

23. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time 72 Hours (AUC0-72): Total HP67.6 Antibody
Description: Area under the plasma concentration-time curve from time zero to the time 72 hours (AUC0-72). Total HP67.6 antibodies analyte was used to determined the AUC0-72 in this outcome measure.
Time Frame: Pre dose, 1, 2, 4, 6, 24 and 72 hours post dose on Cycle 1 Day 1
Population: PK analysis set included all the participants who were treated with GO and contributed at least 1 PK sample. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 48
nanogram*hour/milliliter | 3797 (135)

24. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time 336 Hours (AUC0-336): AC-CL-184538 and CL-184538
Description: Area under the plasma concentration-time curve from time zero to the time 336 hours (AUC0-336). Calicheamicin (conjugated calicheamicin ac-CL-184538 and unconjugated CL-184538) analytes were used to determined the AUC0-336 in this outcome measure.
Time Frame: Pre dose, 2, 4, 6, 72, 192 and 336 hours post dose on Cycle 1 Day 7
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/milliliter
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
picogram*hour/milliliter
  AC-CL-184538: number analyzed (Participants) | 45
  AC-CL-184538 | 461500 (121)
  CL-184538: number analyzed (Participants) | 35
  CL-184538 | 1639 (181)

25. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time 336 Hours (AUC0-336): Total HP67.6 Antibody
Description: Area under the plasma concentration-time curve from time zero to the time 336 hours (AUC0-336). Total HP67.6 antibodies analyte was used to determined the AUC0-336 in this outcome measure.
Time Frame: Pre dose, 2, 4, 6, 72, 192 and 336 hours post dose on Cycle 1 Day 7
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 42
nanogram*hour/milliliter | 26820 (131)

26. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. A treatment emergent AE was defined as an event between first dose of study drug and up to 36 days after the last dose of study drug, that was absent before treatment, or that worsened during the treatment period relative to the pretreatment state. AEs included all serious and non-serious adverse events.
Time Frame: From first dose of study drug up to 36 days after last dose (up to a maximum of 12 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
Participants
  TEAEs | 49
  SAEs | 34

27. Secondary Outcome: Number of Participants With Shift From Grade <=2 at Baseline to Grade 3 or 4 Post-Baseline in Clinical Laboratory Abnormalities- Hematology and Coagulation Parameters
Description: Laboratory parameters included hematological and coagulation parameters. These included activated partial thromboplastin time prolonged, anemia, fibrinogen decreased, hemoglobin increased, international normalized ratio increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, white blood cell decreased. Number of participants with hematological and coagulation abnormalities by grades (as per Common Terminology Criteria for Adverse Events (CTCAE version 4.03) were reported. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: From first dose of study drug up to 36 days after last dose (up to a maximum of 12 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
Participants | 43

28. Secondary Outcome: Number of Participants With Shift From Grade <=2 at Baseline to Grade 3 or 4 Post-Baseline in Clinical Laboratory Abnormalities- Chemistry Parameters
Description: Laboratory parameters included chemistry parameters. These included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatinine increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, and hyponatremia. Number of participants with chemistry test abnormalities by grades (CTCAE version 4.03) were reported. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: From first dose of study drug up to 36 days after last dose (up to a maximum of 12 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
Participants | 18

29. Secondary Outcome: Percentage of Participants With Positive Anti-Drug Antibody (ADA)
Description: Percentage of participants with treatment-induced ADA positive (post baseline-positive only) and treatment-boosted ADA positive (baseline ADA titer that was boosted to a 9-fold or higher level following drug administration) were reported in this outcome measure.
Time Frame: From first dose of study drug up to maximum of 12 months
Population: Immunogenicity analysis set included all participants in the safety analysis set who had at least 1 immunogenicity sample with results.
Measure: Number; unit: percentage of participants
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
percentage of participants
  Treatment-induced ADA Positive | 12.0
  Treatment-boosted ADA Positive | 0.0

30. Secondary Outcome: Percentage of Participants With Positive Neutralizing Antibodies (NAb)
Description: Percentage of participants with either treatment-induced NAb or treatment-boosted NAb were reported.
Time Frame: From first dose of study drug up to maximum of 12 months
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 50
percentage of participants | 2.0

31. Secondary Outcome: Percentage of Participants Who Achieved Complete Remission (CR) and Complete Remission With Incomplete Hematologic Recovery (CRi)
Description: Percentage of participants with first dose of study drug to best overall response with CR and CRi were reported. CR was defined as the disappearance of leukemia indicated by less than (<) 5 percent (%) bone marrow blasts, absence of circulating blasts with auer rods and absence of extramedullary disease, with recovery of hematopoiesis defined by absolute neutrophil count (ANC) greater than or equal to (>=)1000 per microliter (1000/mcL) and platelets >=100,000/mcL. CRi was defined as all CR criteria except residual neutropenia; ANC <1000/mcL or thrombocytopenia and platelet count <100,000/mcL.
Time Frame: From first dose of study drug to 36 days after last dose (maximum up to of 12 months)
Population: Full analysis set included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 51
percentage of participants | 9.8 [3.3 to 21.4]

32. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the start date (first dose) of study treatment to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From the first dose of study treatment to the date of death or date of censored, whichever occurred first (maximum up to 12 months)
Population: Full analysis set included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemtuzumab Ozogamicin (GO)
Number analyzed (Participants) | 51
months | 2.8 [1.7 to 4.2]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 36 days after last dose (up to a maximum of 12 months)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Arm/Group | Gemtuzumab Ozogamicin (GO)
All-Cause Mortality (participants affected / at risk) | 45/50
Serious Adverse Events (participants affected / at risk) | 34/50
Other Adverse Events (participants affected / at risk) | 36/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemtuzumab Ozogamicin (GO) (N=50)
Febrile Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
Vitreous Floaters (Eye disorders) | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 1
Disease Progression (General disorders) | 5
Pyrexia (General disorders) | 3
Multiple Organ Dysfunction Syndrome (General disorders) | 1
Sepsis (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 3
Atypical Pneumonia (Infections and infestations) | 2
Covid-19 Pneumonia (Infections and infestations) | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1
Eye Infection Fungal (Infections and infestations) | 1
Neutropenic Sepsis (Infections and infestations) | 1
Pneumonia Klebsiella (Infections and infestations) | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Capillary Leak Syndrome (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemtuzumab Ozogamicin (GO) (N=50)
Anaemia (Blood and lymphatic system disorders) | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Abdominal Pain Upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Gingival Bleeding (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 3
Chills (General disorders) | 3
Fatigue (General disorders) | 4
Pyrexia (General disorders) | 6
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3
Alanine Aminotransferase Increased (Investigations) | 4
Aspartate Aminotransferase Increased (Investigations) | 5
Gamma-Glutamyltransferase Increased (Investigations) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Headache (Nervous system disorders) | 5
Acute Kidney Injury (Renal and urinary disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT03727750/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03727750/SAP_001.pdf